CLINICAL TRIAL: NCT04146558
Title: A Randomized Open Label Clinical Trial on the Efficacy of an Ayurvedic Treatment Package on Symptom Severity and Quality of Life in Plaque Psoriasis
Brief Title: Ayurvedic Treatment Package in Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Poomulli Neelakandan Namboodiripad Memorial Ayurveda Medical College (Unknown)
Responsible Party: Principal Investigator, Holger Cramer, Professor, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GI012019
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal ayurvedic treatment (Experimental): All possible internal preparations will be administered for a period of 12 months.
  All administered preparations with its dosage and duration will be documented All preparations will be subjected to lab test for clearing heavy metal and pesticide content before the administration
  Interventions: Drug: Individualized internal ayurvedic treatment
- External ayurvedic treatment (Active Comparator): Application of warm external oil (Ayyapala kera tailam) on affected parts twice daily
  Interventions: Other: External ayurvedic treatment

INTERVENTIONS:
Drug: Individualized internal ayurvedic treatment — All possible internal preparations will be administered for a period of 12 months.
  All administered preparations with its dosage and duration will be documented All preparations will be subjected to lab test for clearing heavy metal and pesticide content before the administration
  Arms: Internal ayurvedic treatment
Other: External ayurvedic treatment — Application of warm external oil (Ayyapala kera tailam) on affected parts twice daily
  Arms: External ayurvedic treatment

SUMMARY:
Psoriasis is a chronic, immune-mediated inflammatory skin disease that is associated with substantial impairment of physical and psychological quality of life. The conventional treatment protocols manages the condition but with remissions and relapses which create anxiety in patients. Many of the patients withdraw from active social life as the disease attains chronicity. Several studies are pointing towards a conjoint management strategy incorporating the traditional and alternate medical systems. In this regard, Ayurveda is commonly used by psoriatic patients in India. Considering this fact it is high time to conduct a study to scientifically evaluate the efficacy of Ayurvedic treatment protocol in managing psoriasis as well as its potential to improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis having age 18 years or more
* Patients with moderate-to-severe plaque psoriasis with a PASI score of 12 or higher
* Psoriasis diagnosed 6 months or more before study entry
* Those who are poorly controlled based on physicians assessment with topical treatments, phototherapy, systemic therapy, or a combination of these therapies.
* Participants who have given informed consent.

Exclusion Criteria:

* Participants with other systemic illnesses
* Lactating and pregnant mothers.
* Alcohol dependence/Narcotic dependence /Steroid dependence
* In the judgment of the investigator, unable or unwilling to follow the protocol and instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Psoriasis-specific quality of life | 6 months
  Psoriasis specific DLQI scores

SECONDARY OUTCOMES:
Psoriasis Severity | 3 months
  Psoriasis Area Severity Index (PASI) score
Psoriasis Severity | 6 months
  Psoriasis Area Severity Index (PASI) score
Psoriasis Severity | 12 months
  Psoriasis Area Severity Index (PASI) score
Psoriasis-specific quality of life | 3 months
  Psoriasis specific DLQI scores
Psoriasis-specific quality of life | 12 months
  Psoriasis specific DLQI scores
Adverse events | 3 months
Adverse events | 6 months
Adverse events | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- PNNM Ayurveda College, Shōranūr, Kerala, India

IPD SHARING:
Plan to Share IPD: No